CLINICAL TRIAL: NCT06190925
Title: Clinical Results of Asqelio Trifocal Toric Diffractive Intraocular Lens
Status: Completed | Type: Observational
Sponsor: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASQT042021
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Cataract
Keywords: cataract surgery; intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational prospective clinical study is to learn about the clinical outcomes three months after binocular implantation of Asqelio Trifocal Toric IOL in 30 patients submitted to cataract surgery following standard clinical practice. The main questions it aims to answer are: How rotationally stable is the lens after implantation and how effective is in the correction of refractive astigmatism.

Additionally, the visual performance at different distances will be assessed, as well as the patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to cataract surgery with phacoemulsification with bilateral implantation of Asqelio Trifocal Toric IOL to avoid residual astigmatism
* Patient signing informed consent
* Clear intraocular media, except for cataracts in both eyes prior to surgery
* Monocular potential postoperative visual acuity of 20/25 or better

Exclusion Criteria:

* Corneal astigmatism lower than 0.75D
* Patients who do not provide informed consent
* Patients who do not understand the study procedure
* Previous corneal surgery or trauma
* Irregular cornea (e.g. keratoconus)
* Choroidal hemorrhage
* Microphtalmos
* Severe corneal dystrophy
* Uncontrolled or medically controlled glaucoma
* Clinically significant macular changes
* Concomitant severe eye disease
* Non-age-related cataract
* Severe optic nerve atrophy
* Diabetic retinopathy
* Proliferative diabetic retinopathy
* Amblyopia
* Extremely shallow anterior camera
* Severe chronic uveítis
* Pregnant or nursing
* Rubella
* Mature/dense cataract that makes it difficult to examine the fundus preoperatively.
* Previous retinal detachment
* Concurrent participation in other research with drugs or clinical devices
* Expect to require another eye surgery during the study period

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Regular clinical patients submitted to bilateral conventional cataract surgery using phacoemulsification and implanted with Asqelio Trifocal Toric to eliminate refractive error and presbyopia, also requiring toric correction to avoid residual astigmatism
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Refraction | 3 months after implantation
  Manifest residual refraction after implantation of IOL using subjective refraction methods (D)

SECONDARY OUTCOMES:
Corrected Visual acuity at distance | 3 months after implantation
  Visual acuity at 4m with refractive correction (LogMAR units)
Corrected Visual acuity at intermediate distance | 3 months after implantation
  Visual acuity at 60cm with refractive correction for distance (LogMAR units)
Corrected Visual acuity at near distance | 3 months after implantation
  Visual acuity at 40cm with refractive correction for distance (LogMAR units)
Uncorrected Visual acuity at distance | 3 months after implantation
  Visual acuity at 4m without correction (LogMAR units)
Uncorrected Visual acuity at intermediate distance | 3 months after implantation
  Visual acuity at 60cm without correction (LogMAR units)
Uncorrected Visual acuity at near distance | 3 months after implantation
  Visual acuity at 40cm without correction (LogMAR units)
Binocular defocus curve | 3 months after implantation
  Defocus curve obtained in binocular conditions from +2.00D to -4.00D vergence in 0.5 steps (LogMAR units)
Rotational stability | 3 months after implantation
  Change in IOL axis position determined with slit lamp (degrees)
Contrast sensitivity function | 3 months after implantation
  Contrast sensitivity determined with best correction for distance, under photopic and mesopic conditions, with and without induced glare, using the Clinical Trial Suite (CTS, M&S Technologies, Niles, IL, EEUU) (Log CS units)
Patient reported outcomes - Satisfaction | 3 months after implantation
  Patient reported outcomes obtained by means of the CATQuest9SF questionnaire. 9 items with 4 response options, ranging from 4 for "very great difficulty/very dissatisfied" to 1 for "no difficulty/very satisfied", and a "cannot decide" additional option, which is treated as missing data.
Patient reported outcomes - Visual Symptoms | 3 months after implantation
  Patient reported outcomes on incidence and intensity of visual symptoms obtained by means of a visual symptoms questionnaire. It explores the frequency, intensity and bothersome of 10 different and common visual symptoms. Patients are asked to respond with 4 response options to the frequency of the symptoms, from 1 for "Never" to 4 "Very often", the intensity of the symptom, from 1 for "None" to 4 for "Severe", and the level of bothersome of the symptom, from 1 for "None" to 4 for "A lot".

CONTACTS AND LOCATIONS:
Locations (1):
- OftalVist Alicante, Alicante, Spain